CLINICAL TRIAL: NCT07341685
Title: Comparison of Women With andWithout Primary Dysmenorrhea in Terms of Pain Threshold, Joint Mobility, PhysicalActivity Habit Level, Respiratory Muscle Strength, Menstruation Attitudes andDepressive Symptoms
Brief Title: Comparison of Pain, Physical, and Psychosocial Parameters in Women With and Without Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, Prof.Dr, Izmir Democracy University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Dismenore-35
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Joint Mobility; Physical Activity
MeSH Terms: conditions — Dysmenorrhea; Motor Activity

STUDY DESIGN:
Intervention Model Description: comparing women with primary dysmenorrhea to women without dysmenorrhea. Measurements of pain threshold, joint mobility, physical activity level, respiratory muscle strength, menstrual attitudes, and depressive symptoms are collected in a single visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Dysmenorrhea Group (Other): Female participants diagnosed with primary dysmenorrhea. Pain threshold, joint mobility, physical activity level, respiratory muscle strength, menstrual attitudes, and depressive symptoms are assessed.
  Interventions: Other: Observational Assessment
- Control Group (Other): Female participants without primary dysmenorrhea. Pain threshold, joint mobility, physical activity level, respiratory muscle strength, menstrual attitudes, and depressive symptoms are assessed.
  Interventions: Other: Observational Assessment

INTERVENTIONS:
Other: Observational Assessment — This study does not involve any therapeutic intervention. Participants undergo observational, non-invasive assessments including pain threshold measurement, joint mobility evaluation, physical activity level assessment, respiratory muscle strength testing, menstrual attitude questionnaires, and depressive symptom evaluation.

SUMMARY:
Dysmenorrhea is a common gynecological condition that negatively affects women's physical, psychological, and social well-being. Primary dysmenorrhea (PD) has been associated with reduced pain thresholds in various body regions; however, evidence regarding its relationship with joint mobility, respiratory muscle strength, and psychosocial factors remains limited. In addition, the influence of menstrual attitudes, physical activity habits, and depressive symptoms in women with PD has not been sufficiently explored. Therefore, this study aims to compare women with and without primary dysmenorrhea in terms of pain threshold, joint mobility, physical activity level, respiratory muscle strength, menstrual attitudes, and depressive symptoms. Identifying the parameters affected by PD is essential for developing effective management strategies and may contribute to increased awareness and improved clinical approaches for primary dysmenorrhea.

DETAILED DESCRIPTION:
Dysmenorrhea is a very common gynecological problem among women during the menstrual period and is defined as "painful menstruation." The pain is most commonly experienced in the abdominal and lumbar regions and is typically described as cramping and colicky in nature. Symptoms such as nausea, vomiting, headache, and leg pain may accompany the pain in dysmenorrhea. Dysmenorrhea leads to decreased work productivity, increased tension in social life, and absenteeism from school or work. Dysmenorrhea is classified into two types: primary and secondary.

In women with primary dysmenorrhea (PD), pressure, heat, and electrical pain thresholds in the abdominal, paravertebral, and extremity regions have been shown to decrease during the menstrual phase. However, research on painful pelvic floor regions in women with PD is still in its early stages. There is very limited published data in the literature addressing the optimal management of women with hypermobility and abnormal uterine bleeding. Therefore, it is necessary to determine the relationship between joint mobility and PD. Similarly, no studies have been found examining PD and respiratory muscle strength. On the other hand, positive or negative beliefs related to menstruation and cultural factors may also influence menstrual attitudes. Although a positive relationship between dysmenorrhea and depression is assumed, the evidence remains controversial and limited.

In light of this information, it is of interest to investigate how all these parameters differ in women with PD compared to women without PD. Therefore, the aim of this study is to compare women with and without primary dysmenorrhea in terms of pain threshold, joint mobility, physical activity level, respiratory muscle strength, menstrual attitudes, and depressive symptoms. Identifying which parameters are affected in PD is important for clinicians and researchers in order to determine effective management strategies for primary dysmenorrhea. Thus, it is believed that this study will contribute to the literature by increasing awareness on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 35 years of age
* Have a history of menstrual pain since the first few years after menarche
* Have a menstrual pain intensity of 4 or higher on the VAS in the last 6 months
* Have no pelvic or uterine pathology (e.g., cysts, infections, fibroids)
* Have a regular menstrual cycle
* Be willing to voluntarily participate in the study

Exclusion Criteria:

* Having a neurological, orthopedic, rheumatologic, cardiac, or pulmonary disease
* Being pregnant or suspected of pregnancy
* Having given birth
* Having undergone abdominal, pelvic, or spinal surgery within the past year
* Having a malignant disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only participants experiencing menstrual pain will be included in the study.
Enrollment: 70 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain Threshold | Baseline
  In this study, participants' pressure pain threshold (PPT) will be assessed. A Wagner digital algometer (Wagner Instruments) will be used to evaluate PPT. Participants will be seated on an adjustable chair with their feet fully supported on the floor and their knees flexed at 90 degrees. For PPT assessment, the algometer will be applied perpendicular (90° angle) to the measurement site.
  Measurements will be performed bilaterally at the midpoint of the upper trapezius muscle, 7 cm lateral to the umbilicus on both the right and left sides, at the midpoint of the paravertebral muscles at the level of the fifth lumbar vertebra, and at the midpoint of the thigh. Each measurement will be repeated three times for each site. A minimum interval of 30 seconds will be allowed between repeated measurements at the same site. The value at which pain is first perceived will be recorded, and the mean of the three measurements will be calculated for each site.
Assessment of Joint Mobility | Baseline
  Joint mobility will be assessed using the Beighton criteria. The Beighton score is one of the most commonly used methods for the diagnosis of joint hypermobility. It is a simple scoring system consisting of five maneuvers with a total score of nine points. The first four maneuvers are assessed bilaterally in all extremities, with one point awarded for each successfully performed movement. The fifth maneuver is scored as one point. A total score of at least 4 out of 9 (≥4/9) is required to indicate joint hypermobility.
Assessment of Physical Activity Level | Baseline
  The International Physical Activity Questionnaire (IPAQ) was developed by Craig et al. to assess individuals' physical activity levels. The validity and reliability of the Turkish version were established by Öztürk et al. The questionnaire is available in two forms: long and short. In this study, the short form of the IPAQ will be used. The short form consists of seven items and provides information on the time spent in walking, moderate-intensity, and vigorous-intensity physical activities. Time spent sitting is assessed as a separate item.
  The total score of the short form is calculated by summing the duration (minutes) and frequency (days) of walking, moderate-intensity, and vigorous-intensity activities. Based on these calculations, a score expressed in MET-minutes is obtained. Energy expenditure for physical activities is calculated using MET-minute scores, and participants are classified according to the numerical values derived from the total score.
Assessment of Respiratory Muscle Strength | Baseline
  Respiratory muscle strength will be assessed using the Cosmed Pony FX spirometer. Voluntary measurements of inspiratory and expiratory muscle strength will be performed with a portable mouth pressure device following ATS/ERS guidelines. Maximal static inspiratory pressure (MIP) will be measured during a brief, forceful inspiratory effort from residual volume (Müller maneuver), and maximal static expiratory pressure (MEP) will be measured during maximal expiration at total lung capacity (Valsalva maneuver). Measurements will be repeated until valid values are obtained. If consecutive measurements differ by more than 5% or 5 cmH₂O, the test will be repeated. The highest value will be used for analysis, and reference equations by Evans and Whitelaw will be applied.
Assessment of Menstrual Attitudes | Baseline
  The Menstrual Attitude Questionnaire (MAQ) was developed based on the theory that menstrual attitudes are multidimensional, encompassing both positive and negative perspectives, and that expectations related to physiological and emotional symptoms before or during menstruation may influence behaviors exhibited during this period. The MAQ is a self-administered, easy-to-use questionnaire consisting of 33 items designed to assess positive and negative attitudes toward menstruation.
  The questionnaire includes five subscales: (1) menstruation as a debilitating event (12 items), (2) menstruation as a bothersome event (6 items), (3) menstruation as a natural event (5 items), (4) anticipation/prediction of the onset of menstruation (5 items), and (5) denial of the effects of menstruation (7 items). Items are rated on a 5-point Likert scale ranging from 1 to 5. Higher scores obtained from the subscales indicate a more positive attitude toward menstruation.
Assessment of Depressive Symptoms | Baseline
  Depressive symptoms will be evaluated using the Beck Depression Inventory (BDI). The BDI was developed by combining frequently observed symptoms and attitudes specific to depression, along with commonly exhibited behaviors. The questionnaire has no time limit and can be completed in approximately 10-15 minutes. It consists of 21 symptom categories, with each item rated on a scale from 0 to 3 according to symptom severity.
  Total scores are interpreted as follows: 0-9 indicating no or minimal depression, 10-18 mild depression, 19-29 moderate depression, and 30-63 severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Sezgi Kızılırmak Karataş, Asst.Prof, Principal Investigator — Izmir Democracy University; Büşra Aydın, std., Principal Investigator — Izmir Democracy University; Öykü Dündar, std., Principal Investigator — Izmir Democracy University; Turna Sürmen, std., Principal Investigator — Izmir Democracy University; Nalan Anık, std., Principal Investigator — Izmir Democracy University; Kader İliman, std., Principal Investigator — Izmir Democracy University; Fadıma Kılıç, std., Principal Investigator — Izmir Democracy University

IPD SHARING:
Plan to Share IPD: No